CLINICAL TRIAL: NCT00852696
Title: A Double Blind, Randomized Placebo Controlled Trial of the Perioperative Use of Solifenacin in the Management of Postoperative Overactive Bladder Symptoms in Patients With Mixed Incontinence Undergoing Suburethral Sling Procedures.
Brief Title: Over Active Bladder Patients Having Sling Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left Cleveland Clinic and absolutely no data is available.
Sponsor: Cleveland Clinic Florida (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Hurtado, Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 8867
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Incontinence; Solifenacin; Women; Postoperative
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo Orally 9 weeks once daily.
  Interventions: Other: Placebo
- Solifenacin Group (Experimental): Solifenacin Orally 9 weeks once daily.
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — Solifenacin is used to treat overactive bladder. It works by relaxing the bladder muscles to prevent urgent, frequent, or uncontrolled urination. Take orally once daily for 9 weeks.
  Other Names: Tolterodine Tartrate
  Arms: Solifenacin Group
Other: Placebo — Take orally once daily for 9 weeks.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine whether treatment with anti-muscarinic medications following sub-urethral sling procedures improves overall subjective and objective outcomes in women with mixed incontinence with primary stress symptoms.

DETAILED DESCRIPTION:
Women with mixed incontinence with primary stress symptoms undergoing Sub-Urethral Sling Procedures will be randomized to peri-operative placebo or solifenacin. Subjects in the placebo group will take orally once daily for 9 weeks. Subjects in the Solifenacin group will take orally once daily for 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18
* Patient is appropriate for sub-urethral sling procedure
* Mixed urinary incontinence
* No antimuscarinic therapy for previous 30 days

Exclusion Criteria:

* Uncontrolled narrow angle glaucoma
* Acute cystitis
* Unevaluated hematuria
* Currently using anti-muscarinic therapy
* Unable to complete pre-operative urodynamics
* Contraindication to anti-cholinergic therapy
* Unable or unwilling to complete diaries or quality of life questionaire
* Significant (exteriorized) Pelvic Organ Prolapse

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G W Davila, MD, Principal Investigator — Cleeland Clinic
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment completed in a clinic setting for eligible participants.
Pre-assignment Details: 1 subject enrolled, unknown patient assignment because this study was double blinded. To our knowledge, the participant never started this trial and no data was collected as study was terminated.
Groups:
- Solifenacin Group: Solifenacin Orally 9 weeks once daily and standard of care.
  Solifenacin: Solifenacin is used to treat overactive bladder. It works by relaxing the bladder muscles to prevent urgent, frequent, or uncontrolled urination. Take orally once daily for 9 weeks.
  Principal investigator left the institution, no data is available
- Placebo: Standard of care and placebo
Period: Overall Study
Arm/Group | Solifenacin Group | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 patient enrolled, but no analysis completed as study was double blinded, no data is available. Baseline data was not collected.
Arm/Group | Solifenacin Group
Number analyzed (Participants) | 0
Age, Continuous [unit: 0]
Sex: Female, Male
Principal investigator left the institution, no data is available.

OUTCOME MEASURES:

1. Primary Outcome: To Determine Whether Treatment With Anti-muscarinic Medications Following Sub-urethral Sling Procedures Improves Overall Subjective and Objective Outcomes in Women With Mixed Incontinence With Primary Stress Symptoms.
Description: Women with mixed incontinence with primary stress symptoms undergoing Sub-Urethral Sling Procedures will be randomized to peri-operative placebo or solifenacin. Subjects in the placebo group will take orally once daily for 9 weeks. Subjects in the Solifenacin group will take orally once daily for 9 weeks.
Time Frame: 9 weeks
Population: Principal investigator left the institution, no data is available.
  1 subject enrolled, unknown patient assignment because this study was double blinded. Data was never collected for this study.
Arm/Group | Solifenacin Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 Weeks Principal investigator left the institution, no data is available
Description: Principal investigator left the institution, no data is available
Groups:
- Solifenacin Group: 1 subject enrolled, unknown patient assignment because this study was double blinded.
Arm/Group | Solifenacin Group
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes